CLINICAL TRIAL: NCT04381351
Title: The Role of Noncoding RNAs in COVID-19 and COVID-19 Associated Acute Kidney Injury (MiRCOVID)
Brief Title: Noncoding RNAs in COVID-19 and COVID-19 Related Kidney Dysfunction
Acronym: MiRCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, Principal Investigator, Heinrich-Heine University, Duesseldorf
Other Study IDs: 1
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: acute kidney injury (AKI); organ dysfunction
MeSH Terms: conditions — COVID-19; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, critically ill patients with highly suspected or confirmed COVID-19 will be included. Main goal is the identification of noncoding RNAs in COVID-19 associated organ dysfunction with an emphasis on acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19

Exclusion Criteria:

* kidney transplantation
* eGFR < 30 ml/Min
* dialysis within last 90 days
* chronic dialysis
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients with critical illness on ICU.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
predicitive value of noncoding RNAs in COVID-19 associated organ dysfunction | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Anästhesiologie, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided